CLINICAL TRIAL: NCT00349427
Title: A Randomized, Double-Blind, Placebo-Control, Clinical Evaluation of Insulin Plus Rosiglitazone Compared to Insulin Plus Placebo for 24 Weeks in Subjects With Type 2 Diabetes Mellitus Who Are Inadequately Controlled On Insulin
Brief Title: A Study Of Rosiglitazone Plus Insulin To Treat Type 2 Diabetes Mellitus Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AVD102209
Record Dates: First submitted 2006-07-06; First posted 2006-07-07 (Estimated); Last update posted 2012-06-04 (Estimated); Status verified 2011-02

CONDITIONS: Type 2 Diabetes Mellitus; Diabetes Mellitus, Type 2
Keywords: Insulin; BRL49653 /rosiglitazone; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance | interventions — Rosiglitazone; Insulin

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Rosiglitazone (Experimental): 4mg
  Interventions: Drug: Rosiglitazone 4 mg
- Rosiglitazone placebo (Placebo Comparator): 4mg
  Interventions: Drug: Rosiglitazone 4 mg

INTERVENTIONS:
Drug: Rosiglitazone 4 mg
  Other Names: Insulin

SUMMARY:
This study is designed to demonstrate that addition of rosiglitazone (4mg) to insulin in Type 2 diabetes mellitus subjects who have not achieved glycemic goals on insulin injections alone is efficacious in terms of improving glycemic control.

ELIGIBILITY:
Inclusion:

* Patients with type 2 Diabetes mellitus on a minimum dose of 30 units/day insulin monotherapy continuously for at least 8 weeks
* If Patients are taking another oral antidiabetic agent may stop their oral agent and adjust their insulin dose properly over 8 weeks prior to screening if they are asked by doctor who considers him/her suitable for study in all other respects, and the HbA1c level>7.5%.

Exclusion:

* Fasting plasma glucose >13 mmol/L at screening
* Ongoing edema or history of peripheral edema requiring pharmacological treatment within 12 months
* Drug abuse
* Women pregnant or lactating
* Use any rosiglitazone like drug in 3 months
* Use more than one oral antidiabetic agent in 2 months
* Uncontrolled hypertension
* Chronic heart failure
* Anemia

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2005-10

PRIMARY OUTCOMES:
glycemic control at treatment 24-week measured by HbA1c (Glycosylated hemoglobin) | 24 weeks

SECONDARY OUTCOMES:
glycemic control at treatment 24-week measured by fasting plasma glucose and daily insulin dose, proportion of subjects who reduce total daily insulin dose after treatment of 8, 16, and 24 weeks | 8, 16, and 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (5):
- China (5):
  - GSK Investigational Site, Nanjing, Jiangsu
  - GSK Investigational Site, Xian, Shanxi
  - GSK Investigational Site, Beijing
  - GSK Investigational Site, Shanghai
  - GSK Investigational Site, Tianjin